CLINICAL TRIAL: NCT05118438
Title: Development of a Health Promotion Nursing Intervention for Post-traumatic Stress Women Based on Swanson's Theory of Caring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Y-2019-0153
Record Dates: First submitted 2021-10-29; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Women Who Have Experienced Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing intervention (Experimental): The recruited participants were clients of a self-sufficiency support center for sexually exploited women located in South Korea, recruited through snowball sampling after obtaining permission from the director of the support center.
  Interventions: Other: Health Promotion Nursing Intervention

INTERVENTIONS:
Other: Health Promotion Nursing Intervention — A one-on-one program was conducted over six sessions, with each session ranging from 60 to 120 minutes. The caring program for health promotion included the following concepts: understanding the self; sharing traumatic events and negative emotions; re-framing the meaning of traumatic events; identifying thoughts and physical and emotional responses; developing health-promoting activities; and maintaining a positive attitude during the process of change .

SUMMARY:
Objectives: We aimed to (1) develop a caring program for health promotion among women who experienced trauma and (2) evaluate its effect on post-traumatic stress, depression, health-promoting behaviors, and self-esteem.

Methods: We conducted a quasi-experimental study using a group pre-test/post-test design. Data were collected from 14 women recruited from a self-sufficiency support center for sexually exploited women who experienced trauma, during December 2019-May 2020. Participants were assessed at pre-test, post-test, and at a one-month follow-up. We analyzed changes in outcome variables over time using repeated-measures analysis of variance and paired t-tests.

ELIGIBILITY:
Inclusion Criteria:

1. women aged over 18 years who had experienced a traumatic event, and
2. a PTS score of 64 or lower on the PTSD checklist for DSM-5 (PCL-5) developed by Weathers et al. (1993), revised by Weathers et al. (2013), and translated into Korean by Kim et al. (2017).

Exclusion Criteria:

1. presence of psychiatric conditions with hallucinations and delusions, and
2. diagnosis of an intellectual disability that would make understanding the intervention procedure difficult. Although a standard cut-off was not present in the PCL-5, women who exceeded 80% (64 points) of the total score were excluded to rule out high-risk women with severe trauma.

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Our study targeted sexually exploited women by family member, previous boyfriends, and strangers.
Enrollment: 14 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
post-traumatic stress | one month after the intervention
  PTS was measured using the PCL-5, which was developed by Weathers et al. (1993), revised by Weathers et al. (2013) as per the revised PTSD definition in the DSM-5, and translated into Korean by Kim et al. (2017). The Korean version of the PCL for the DSM-5 (PCL-5-K) contains 20 items, and each scored from 0 (not at all) to 4 (extremely). The score depended on the severity of the symptom caused by stress related to traumatic events during the past month. Possible scores ranged from 0 to 80, with a score of 37 or above indicating a PTSD diagnosis, and higher scores suggesting severe PTSD symptoms (Kim et al., 2017). Cronbach's alpha coefficient for the PCL-5-K was .97 among Korean veterans of the Vietnam War (Kim et al., 2017) and .89 in the current study.
depression | one month after the intervention
  Depression was assessed using the Center for Epidemiologic Studies Depression Scale (CES-D), developed by Radloff (1977), and translated into Korean by Chon and Rhee (1992). The Korean version of the CES-D contains 20 items rated on a 4-point Likert scale (0 = rarely or never; to 3 = all the time), according to how respondents felt during the past week. Possible scores ranged from 0 to 60, with a score of 16 or above indicating depressive symptoms, and higher scores indicating higher levels of depression (Radloff, 1977). Cronbach's alpha coefficient for the Korean CES-D was .89 among Korean adults (Chon & Rhee, 1992) and .78 in our study.
health-promoting behaviors | one month after the intervention
  Health-promoting behaviors were measured using the Health Promoting Lifestyle Profile-II (HPLP-II), developed by Walker et al. (1995) and translated into Korean by Yun and Kim (1999). The Korean version of the HPLP-II comprises 52 items under six subscales: health responsibility (scores ranging from 9-36), physical activity (scores ranging from 8-32), nutrition (scores ranging from 9-36), spiritual growth (scores ranging from 9-36), interpersonal relations (scores ranging from 9-36), and stress management (scores ranging from 8-32). It was rated on a 4-point Likert scale (1=never, 2=sometimes, 3=often, 4=routinely). Possible scores ranged from 52 to 208, with higher scores indicating higher levels of health-promoting behaviors. Cronbach's alpha coefficients were .78, .87, .69, .77, .81, and .73 for health responsibility, physical activity, nutrition, spiritual growth, interpersonal relations, and stress management, respectively.
self-esteem | one month after the intervention
  Self-esteem was assessed using the Rosenberg Self Esteem Scale (RSES), developed by Rosenberg (1965), and translated into Korean by Bae et al. (2014). The Korean version of the RSES (K-RSES) comprises ten items rated on a 4-point Likert scale, ranging from strongly agree to strongly disagree. Possible scores ranged from 10 to 40, with higher scores indicating higher self-esteem. Cronbach's alpha coefficient for the K-RSES was .90 among Korean adults (Bae et al., 2014) and .90 in our study.

CONTACTS AND LOCATIONS:
Overall Officials: Go-Un Kim, Principal Investigator — College of Nursing and Mo-Im Kim Nursing Research Institute, Yonsei University
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No